CLINICAL TRIAL: NCT02218723
Title: An Open-label, Randomised, Cross-over, Single Dose Study in Healthy Volunteers to Evaluate the Unit Dose Dry Powder Inhaler (UD-DPI) With Four Different Formulations for the Delivery of Fluticasone Furoate and to Compare the Pharmacokinetic Profile With the Fluticasone Furorate ELLIPTA Presentation
Brief Title: Pharmacokinetic Profile of Four Formulations of Fluticasone Furoate (FF) Using Unit Dose Dry Powder Inhaler (UD-DPI) Compared With FF ELLIPTA® Presentation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200939
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Asthma
Keywords: healthy volunteer; Asthma; inhaled corticosteroid; UD-DPI; ELLIPTA DPI; Fluticasone furoate
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Sequence ABECD (Active Comparator): Subject will be administered treatment in sequence ABECD. Where, A: a single dose of FF [100 microgram (mcg) per blister from 0.6% blend] delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; B: a single dose of FF (80mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 320mcg; C: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; D: a single dose of FF (140mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 560mcg; E: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the ELLIPTA DPI by inhalation of 4 Blisters giving a total dose of 400mcg
  Interventions: Drug: FF UD-DPI; Drug: FF ELLIPTA DPI
- Sequence BCADE (Active Comparator): Subject will be administered treatment in sequence BCADE. Where, A: a single dose of FF (100mcg per blister from 0.6% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; B: a single dose of FF (80mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 320mcg; C: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; D: a single dose of FF (140mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 560mcg; E: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the ELLIPTA DPI by inhalation of 4 Blisters giving a total dose of 400mcg
  Interventions: Drug: FF UD-DPI; Drug: FF ELLIPTA DPI
- Sequence CDBEA (Active Comparator): Subject will be administered treatment in sequence CDBEA. Where, A: a single dose of FF (100mcg per blister from 0.6% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; B: a single dose of FF (80mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 320mcg; C: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; D: a single dose of FF (140mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 560mcg; E: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the ELLIPTA DPI by inhalation of 4 Blisters giving a total dose of 400mcg
  Interventions: Drug: FF UD-DPI; Drug: FF ELLIPTA DPI
- Sequence DECAB (Active Comparator): Subject will be administered treatment in sequence DECAB. Where, A: a single dose of FF (100mcg per blister from 0.6% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; B: a single dose of FF (80mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 320mcg; C: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; D: a single dose of FF (140mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 560mcg; E: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the ELLIPTA DPI by inhalation of 4 Blisters giving a total dose of 400mcg
  Interventions: Drug: FF UD-DPI; Drug: FF ELLIPTA DPI
- Sequence EADBC (Active Comparator): Subject will be administered treatment in sequence EADBC. Where, A: a single dose of FF (100mcg per blister from 0.6% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; B: a single dose of FF (80mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 320mcg; C: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; D: a single dose of FF (140mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 560mcg; E: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the ELLIPTA DPI by inhalation of 4 Blisters giving a total dose of 400mcg
  Interventions: Drug: FF UD-DPI; Drug: FF ELLIPTA DPI
- Sequence DCEBA (Active Comparator): Subject will be administered treatment in sequence DCEBA. Where, A: a single dose of FF (100mcg per blister from 0.6% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; B: a single dose of FF (80mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 320mcg; C: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; D: a single dose of FF (140mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 560mcg; E: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the ELLIPTA DPI by inhalation of 4 Blisters giving a total dose of 400mcg
  Interventions: Drug: FF UD-DPI; Drug: FF ELLIPTA DPI
- Sequence EDACB (Active Comparator): Subject will be administered treatment in sequence EDACB. Where, A: a single dose of FF (100mcg per blister from 0.6% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; B: a single dose of FF (80mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 320mcg; C: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; D: a single dose of FF (140mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 560mcg; E: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the ELLIPTA DPI by inhalation of 4 Blisters giving a total dose of 400mcg
  Interventions: Drug: FF UD-DPI; Drug: FF ELLIPTA DPI
- Sequence AEBDC (Active Comparator): Subject will be administered treatment in sequence AEBDC. Where, A: a single dose of FF (100mcg per blister from 0.6% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; B: a single dose of FF (80mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 320mcg; C: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; D: a single dose of FF (140mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 560mcg; E: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the ELLIPTA DPI by inhalation of 4 Blisters giving a total dose of 400mcg
  Interventions: Drug: FF UD-DPI; Drug: FF ELLIPTA DPI
- Sequence BACED (Active Comparator): Subject will be administered treatment in sequence BACED. Where, A: a single dose of FF (100mcg per blister from 0.6% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; B: a single dose of FF (80mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 320mcg; C: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; D: a single dose of FF (140mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 560mcg; E: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the ELLIPTA DPI by inhalation of 4 Blisters giving a total dose of 400mcg
  Interventions: Drug: FF UD-DPI; Drug: FF ELLIPTA DPI
- Sequence CBDAE (Active Comparator): Subject will be administered treatment in sequence CBDAE. Where, A: a single dose of FF (100mcg per blister from 0.6% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; B: a single dose of FF (80mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 320mcg; C: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 400mcg; D: a single dose of FF (140mcg per Blister from a 0.8% blend) delivered via the UD-DPI by inhalation of 4 Blisters giving a total dose of 560mcg; E: a single dose of FF (100mcg per Blister from a 0.8% blend) delivered via the ELLIPTA DPI by inhalation of 4 Blisters giving a total dose of 400mcg
  Interventions: Drug: FF UD-DPI; Drug: FF ELLIPTA DPI

INTERVENTIONS:
Drug: FF UD-DPI — A blister containing a small quantity of powder comprising of a blend of FF (micronised) and excipient(s) will be administered using UD-DPI. It is available in following dosages: 80mcg/Blister (0.8% Blend); 100mcg/Blister (0.8% Blend); 140mcg/Blister (0.8% Blend); 100mcg/Blister (0.6% Blend)
Drug: FF ELLIPTA DPI — A blister strip contained within the ELLIPTA device. Each blister contains a small quantity of powder comprising of a blend of FF and excipient(s) in dose 100mcg/Blister (0.8% Blend)

SUMMARY:
This is an open-label, five- period, cross-over, randomized, single dose, single centre study in healthy subjects. This is the second clinical study for the UD-DPI. This study will ascertain whether the Pharmacokinetics (PK) systemic exposure [in terms of area under the plasma concentration-time curve (AUC) and maximum observed plasma concentration (Cmax)] of FF delivered via the UD-DPI is comparable to the systemic exposure of FF delivered via the ELLIPTA Dry Powder Inhaler (DPI). For this reason four treatment doses consisting of three dose strengths and 2 percentage blends will be assessed when delivered via the UD-DPI. This study is designed to compare the pharmacokinetic profile of various doses and blends of FF administered via UD-DPI and relative to FF administered via ELLIPTA DPI. Subjects will be screened 28 days prior to study initiation. During each treatment period, subjects will be at study site from evening prior to dosing until completion of the 48 hour post-dose PK sample collection on Day 3. Minimum 7 days washout will be between treatments after completion of all five treatments and the follow-up visit will be conducted 7-14 days post last dose. Duration of study is 13 weeks. ELLIPTA is a registered trademark of the GSK group of companies.

ELIGIBILITY:
Inclusion Criteria:

* AGE- Between 18 and 65 years of age inclusive, at the time of signing the informed consent
* TYPE OF SUBJECT AND DIAGNOSIS INCLUDING DISEASE SEVERITY
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, and laboratory tests.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* WEIGHT-Body Weight >= 50 kilogram and BMI within the range 19.0 - 34.0 kilogram per square metre (inclusive)
* SEX
* Male,
* Female subject : is eligible to participate if she is not pregnant [as confirmed by a negative serum human chorionic gonadotrophin (hCG) test at screening or urine hCG prior to dosing], not lactating, and at least one of the following conditions applies:
* Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy
* Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
* Reproductive potential and agrees to follow one of the options listed below in the GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication and until completion of the follow-up visit.
* GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP)
* This list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis.
* Contraceptive subdermal implant that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label
* Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label
* Oral Contraceptive, either combined or progestogen alone
* Injectable progestogen
* Contraceptive vaginal ring
* Percutaneous contraceptive patches
* Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject
* These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* INFORMED CONSENT Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in protocol.
* OTHER
* Capable of using the UD-DPI and the ELLIPTA DPI adequately after training
* Subjects who are current non-smokers, who have not used any tobacco products in the 6 month period preceding the screening visit, and have a pack history of <= 5 pack years.
* Number of pack years = (number of cigarettes per day/20) x number of years smoked

Exclusion Criteria:

* CONCURRENT CONDITIONS/MEDICAL HISTORY (INCLUDES LIVER FUNCTION AND QTc INTERVAL
* Alanine transaminase (ALT) and bilirubin >1.5x Upper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Clinically significant abnormal ECG finding. Significant is defined as any finding that, in the opinion of the investigator, would put the safety of the subject at risk through participation.
* CONCOMITANT MEDICATIONS
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, or use of St. John's Wort within 14 days prior to the first dose of study medication. By exception, the volunteer may take paracetamol (<=2 grams/day) any time during the study. However, the Investigator and GSK study team can review medication on a case by case basis to determine if its use would compromise subject safety or interfere with the study procedures or data interpretation
* RELEVANT HABITS
* History of regular alcohol consumption within 2 months of the study defined as:
* For Australian sites: An average weekly intake of >21 units for males or >14 units for females. One unit (= standard drink) is equivalent to 10 g of alcohol: 270ml of full strength beer (4.8%), 375mL of mid strength beer (3.5%), 470mL of light beer (2.7%), 250mL pre-mix full strength spirit (5%), 100mL of wine (13.5%) and 30mL of spirit (40%).
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* An unwillingness to abstain from strenuous exercise starting 72 hours prior to each dosing day
* An unwillingness to abstain from caffeine- and xantheine- containing products for 24 hours prior to dosing.
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* CONTRAINDICATIONS
* Drug Allergy:
* Any immediate or delayed hypersensitivity reaction to a corticosteroid (i.e., intranasal, inhaled, systemic therapy).
* Known or suspected sensitivity to the constituents of the DPI or (i.e., lactose or magnesium stearate).
* Milk Protein Allergy: History of severe milk protein allergy.
* History of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* The subject has taken systemic, oral or depot corticosteroids less than 12 weeks before the screening visit.
* The subject has taken inhaled, intranasal or topical steroids less than 4 weeks before the screening visit.
* DIAGNOSTIC ASSESSMENTS AND OTHER CRITERIA
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. . For potent immunosuppressive agents, subjects with presence of hepatitis B core antibody (HBcAb) should also be excluded.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 millilitre (mL) within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* The subject has a history of breathing problems in adult life (e.g. history of asthmatic symptomatology). Screening lung function tests will be performed to confirm normal lung function parameters Forced Expiratory Volume in 1 Second (FEV1) >=85% predicted and FEV1/ Forced Vital capacity (FVC) ratio >=0.7).
* Subjects who have suffered a lower respiratory tract infection within 4 weeks of the screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2014-12-19 (Actual); Study Completion 2014-12-19 (Actual)

PRIMARY OUTCOMES:
AUC from time zero (pre-dose) to 24 hours (hr) (AUC [0-24hr]) and/ or AUC from time zero extrapolated to infinite time (AUC [0-infinity]) and/ or AUC from time zero to last time of quantifiable concentration (AUC [0-t]) | Day 1, Day 2 and Day3 of each period
  AUC (0-24h) and/or AUC(0-t) and/or AUC(0- infinity) will be measured at predose, 5 minutes (min), 10 min, 20 min, 30 min and 45 min, 1 hr, 1.5 hr, 2 hr, 3 hr,4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr, 24 hr, 36 hr and 48 hr

SECONDARY OUTCOMES:
Cmax | Day 1, Day 2 and Day3 of each period
  Cmax will be measured at predose, 5 min, 10 min, 20 min, 30 min and 45 min, 1 hr, 1.5 hr, 2 hr, 3 hr,4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr, 24 hr, 36 hr and 48 hr
Time to Cmax (tmax) | Day 1, Day 2 and Day3 of each period
  Tmax will be measured at predose, 5 min, 10 min, 20 min, 30 min and 45 min, 1 hr, 1.5 hr, 2 hr, 3 hr,4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr, 24 hr, 36 hr and 48 hr
Safety as assessed by adverse events (AE) | Up to Week 13
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Safety as assessed by 12 Lead Electrocardiogram (ECG) Parameters | Day 1 in each period
  Single 12-lead ECGs will be measured in a semi-supine position at each timepoint during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT duration corrected
Safety as assessed by Vital signs | Day 1, Day 3 in each period
  Vital signs include temperature, systolic and diastolic blood pressure, heart rate

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Australia (2):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: Results for study 200939 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200939?search=study&study_ids=200939#rs